CLINICAL TRIAL: NCT00720499
Title: Randomised, Double-blind, Cross-over Study to Assess the Efficacy and Safety of 4 Weeks of Once Daily Treatment of 2 Doses of Orally Inhaled BI 1744 CL, Each in Fixed Dose Combination (FDC) With 5 Microgram Tiotropium Bromide (Delivered by the Respimat® Inhaler) in Patients With COPD
Brief Title: Efficacy and Safety of 4 Weeks of Treatment With Orally Inhaled BI1744/Tiotropium Bromide in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.9; EudtaCT No: 2008-000562-23
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BI 1744 CL low dose+tiotropium bromide (Experimental): BI 1744 CL low dose plus tiotropium bromide fixed dose combination; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
  Interventions: Drug: BI 1744 CL plus tiotropium bromide; Device: Respimat® Inhaler
- BI 1744 CL medium dose+tiotropium bromide (Experimental): BI 1744 CL medium dose plus tiotropium bromide fixed dose combination; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
  Interventions: Drug: BI 1744 CL plus tiotropium bromide; Device: Respimat® Inhaler

INTERVENTIONS:
Drug: BI 1744 CL plus tiotropium bromide — BI 1744 CL plus tiotropium bromide fixed dose combination; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
Device: Respimat® Inhaler

SUMMARY:
The primary objective of this study is to determine the optimum dose(s) of BI 1744 CL administered with 5 microgram tiotropium bromide solution for inhalation, delivered by the Respimat® inhaler, once daily for four weeks in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable airway obstruction with a post-bronchodilator FEV1 >= 30% of predicted normal and <80% of predicted normal and a post-bronchodilator FEV1 / FVC <70% at Visit 1
3. Male or female patients, 40 years of age or older
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years
5. Patients must be able to perform technically acceptable pulmonary function tests and PEF measurements, and must be able to maintain records (Patient Daily e-Diary) during the study period as required in the protocol
6. Patients must be able to inhale medication in a competent manner from the Respimat inhaler and from a metered dose inhaler (MDI).
7. additional inclusion criteria apply.

Exclusion Criteria:

1. Patients with a significant disease other than COPD
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis;
3. Patients with a history of asthma or a total blood eosinophil count >= 600/mm3.
4. Patients with any of the following conditions:a diagnosis of thyrotoxicosis, a diagnosis of paroxysmal tachycardia (>100 beats per minute), a marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTcF* interval > 450 ms), a history of additional risk factors for Torsade de Pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT Syndrome)
5. Patients with any of the following conditions:a history of myocardial infarction within 1 year of screening visit (Visit 1), a diagnosis of clinically relevant cardiac arrhythmia, known active tuberculosis, a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years, a history of life-threatening pulmonary obstruction, a history of cystic fibrosis, clinically evident bronchiectasis, a history of significant alcohol or drug abuse
6. Patients who have undergone thoracotomy with pulmonary resection
7. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits.
8. Pregnant or nursing women
9. Women of childbearing potential not using two effective method of birth control (one barrier and one non-barrier). Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years
10. Patients who have previously been randomized in this study or are currently participating in another study
11. Patients who are unable to comply with pulmonary medication restrictions prior to randomization
12. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit
13. additional exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (24):
- United States (5):
  - 1237.9.00152 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1237.9.00155 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1237.9.00151 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1237.9.00154 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1237.9.00153 Boehringer Ingelheim Investigational Site, Spokane, Washington
- Belgium (5):
  - 1237.9.03253 Boehringer Ingelheim Investigational Site, Brussels
  - 1237.9.03255 Boehringer Ingelheim Investigational Site, Brussels
  - 1237.9.03254 Boehringer Ingelheim Investigational Site, Edegem
  - 1237.9.03251 Boehringer Ingelheim Investigational Site, Ghent
  - 1237.9.03252 Boehringer Ingelheim Investigational Site, Leuven
- Canada (5):
  - 1237.9.00255 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1237.9.00251 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.9.00252 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.9.00254 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.9.00253 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
- Germany (9):
  - 1237.9.04952 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.9.04953 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.9.04954 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.9.04955 Boehringer Ingelheim Investigational Site, Bruchsal
  - 1237.9.04959 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 1237.9.04960 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1237.9.04958 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.9.04951 Boehringer Ingelheim Investigational Site, Tübingen
  - 1237.9.04956 Boehringer Ingelheim Investigational Site, Wiesloch

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, 2-way cross-over trial. 141 patients were randomized to one of 2 treatments sequences and treated. It was a double-blind trial in which each treatment period lasted 4 weeks. During the 2 week pre-treatment run-in and during the 2 week washout between treatment periods, patients received open-label tiotropium 5µg.
Groups:
- Tio+Olo 5/2µg / Tio+Olo5/5µg: Patients received fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol (BI1744) 2 µg followed by fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol (BI1744) 5 µg.
  Both treatments were administered once daily in the morning via the respimat inhaler.
- Tio+Olo5/5µg / Tio+Olo5/2µg: Patients received fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol (BI1744) 5 µg followed by fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol (BI1744) 2 µg.
  Both treatments were administered once daily in the morning via the respimat inhaler.
Period: Treatment Period 1 (4 Weeks)
Arm/Group | Tio+Olo 5/2µg / Tio+Olo5/5µg | Tio+Olo5/5µg / Tio+Olo5/2µg
Started | 69 | 72
Completed | 66 | 70
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 1 | 2
Period: Washout Period (2 Weeks)
Arm/Group | Tio+Olo 5/2µg / Tio+Olo5/5µg | Tio+Olo5/5µg / Tio+Olo5/2µg
Started | 66 | 70
Completed | 66 | 70
Not Completed | 0 | 0
Period: Treatment Period 2 (4 Weeks)
Arm/Group | Tio+Olo 5/2µg / Tio+Olo5/5µg | Tio+Olo5/5µg / Tio+Olo5/2µg
Started | 66 | 70
Completed | 64 | 67
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: A randomised, double-blind, 2-way cross-over study. The two treatment periods were separated by a wash-out period of 14 days during which they received open-label Tiotropium 5 mcg. The 2 treatments, administered once daily in the morning via the respimat inhaler, were :
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 2 µg
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg
Arm/Group | Overall Study
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.67 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 93

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) Response [L] After Four Weeks of Treatment.
Description: Trough FEV1 was defined as the mean of the 2 FEV1 values at the end of the dosing interval, 24 hours post-drug administration.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1 hour (h), 10 minutes (min) before drug administration and 5min, 30min, 1h, 2h, 3h, 4h, 5h, 6h after drug administration on day 29
Population: Full analysis Set (FAS) which included all randomized patients who received at least one dose of study medication and had baseline data and Washout Period for at least 1 efficacy endpoint for each treatment period.
Measure: Mean (Standard Error); unit: Litres
Groups:
- Olo 2 µg + Tio 5 µg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 2 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 1.0 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Olo 5 µg + Tio5 µg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres | 0.057 (0.013) | 0.055 (0.013)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.8937, ANCOVA; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.035 to 0.031], Standard Error of Mean 0.017 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

2. Secondary Outcome: Trough FEV1 Response [L] After 2 Weeks of Treatment
Description: Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h after drug administration on day 15
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres | 0.037 (0.015) | 0.059 (0.015)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.2425, ANCOVA; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.015 to 0.061], Standard Error of Mean 0.019 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

3. Secondary Outcome: Individual FEV1 Measurements
Description: Individual FEV1 measurements [L] at each time point on Day 29.
  The presented means are adjusted.
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h, 4h, 5h, 6h after drug administration on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres
  -1:00 | 1.426 (0.013) | 1.417 (0.013)
  -0:10 | 1.434 (0.014) | 1.438 (0.014)
  0:05 | 1.497 (0.014) | 1.498 (0.014)
  0:30 | 1.541 (0.012) | 1.534 (0.012)
  1:00 | 1.570 (0.012) | 1.570 (0.012)
  2:00 | 1.617 (0.012) | 1.614 (0.012)
  3:00 | 1.601 (0.015) | 1.606 (0.015)
  4:00 | 1.582 (0.016) | 1.606 (0.016)
  5:00 | 1.571 (0.013) | 1.570 (0.014)
  6:00 | 1.547 (0.013) | 1.551 (0.013)

4. Secondary Outcome: FEV1 AUC 0-3h, Response
Description: FEV1 Area Under the Curve (AUC) 0-3h, response [L] on days 1, 15 and 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h after drug administration on days 1, 15 and 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres
  Day 1 | 0.168 (0.006) | 0.173 (0.006)
  Day 15 | 0.174 (0.012) | 0.194 (0.012)
  Day 29 | 0.201 (0.011) | 0.200 (0.011)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Test Day 1. Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.5198, ANCOVA; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.010 to 0.021], Standard Error of Mean 0.008 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Test Day 15. Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.2110, ANCOVA; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.011 to 0.051], Standard Error of Mean 0.016 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 3: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Test day 29. Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.9368, ANCOVA; Mean Difference (Final Values) = -0.001, 95% CI 2-sided [-0.029 to 0.027], Standard Error of Mean 0.014 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

5. Secondary Outcome: FEV1 Peak 0-3h Response
Description: FEV1 peak value over the time from 0 to 3 hours (peak 0-3h) response [L] on days 1, 15 and 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h after drug administration on days 1, 15 and 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres
  Day 1 | 0.269 (0.008) | 0.262 (0.008)
  Day 15 | 0.257 (0.014) | 0.279 (0.015)
  Day 29 | 0.288 (0.014) | 0.294 (0.014)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5339, ANCOVA; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.027 to 0.014], Standard Error of Mean 0.010 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.2408, ANCOVA; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.015 to 0.058], Standard Error of Mean 0.019 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 3: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.7139, ANCOVA; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.029 to 0.042], Standard Error of Mean 0.018 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

6. Secondary Outcome: FEV1, AUC (0-6h) Response
Description: FEV1, AUC (0-6h) response [L] on day 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h, 4h, 5h, 6h after drug administration on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres | 0.202 (0.012) | 0.206 (0.012)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.7906, ANCOVA; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.026 to 0.034], Standard Error of Mean 0.015 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

7. Secondary Outcome: FEV1 (Unsupervised) AUC (6-12h) Response
Description: FEV1 (unsupervised) AUC (6-12h) response [L] on day 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 6 hours (h), 9h and 12h after drug administration on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 130 | 132
Litres | 0.106 (0.029) | 0.114 (0.029)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.8473, ANCOVA; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.067 to 0.082], Standard Error of Mean 0.038 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

8. Secondary Outcome: Trough FVC Response
Description: Trough Forced Vital Capacity (FVC) response [L] on days 15 and 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h after drug administration on day 15, in addition 4h, 5h, 6h after drug administration on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres
  Day 15 | 0.072 (0.024) | 0.104 (0.025)
  Day 29 | 0.066 (0.022) | 0.076 (0.023)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.2944, ANCOVA; Mean Difference (Final Values) = 0.032, 95% CI 2-sided [-0.029 to 0.094], Standard Error of Mean 0.031 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.7180, ANCOVA; Mean Difference (Final Values) = 0.010, 95% CI 2-sided [-0.046 to 0.066], Standard Error of Mean 0.028 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

9. Secondary Outcome: Individual FVC Measurements
Description: Individual FVC measurements [L] at each time point
  The categories correspond to the planned times for FVC measurements on Day 29.
  The presented means are adjusted.
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h, 4h, 5h, 6h after drug administration on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres
  -1:00 | 2.894 (0.023) | 2.899 (0.024)
  -0:10 | 2.892 (0.024) | 2.907 (0.024)
  0:05 | 3.009 (0.024) | 3.032 (0.025)
  0:30 | 3.067 (0.023) | 3.083 (0.024)
  1:00 | 3.093 (0.023) | 3.112 (0.023)
  2:00 | 3.154 (0.023) | 3.189 (0.023)
  3:00 | 3.147 (0.037) | 3.201 (0.038)
  4:00 | 3.143 (0.039) | 3.204 (0.040)
  5:00 | 3.109 (0.025) | 3.131 (0.025)
  6:00 | 3.061 (0.023) | 3.083 (0.023)

10. Secondary Outcome: FVC AUC (0-3h) Response
Description: FVC AUC (0-3h) response [L] on days 1, 15 and 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h after drug administration on days 1, 15 and 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres
  Day 1 | 0.273 (0.012) | 0.275 (0.012)
  Day 15 | 0.271 (0.020) | 0.308 (0.021)
  Day 29 | 0.275 (0.021) | 0.303 (0.022)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9384, ANCOVA; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.029 to 0.032], Standard Error of Mean 0.015 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.1583, ANCOVA; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [-0.014 to 0.088], Standard Error of Mean 0.026 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 3: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.2914, ANCOVA; Mean Difference (Final Values) = 0.029, 95% CI 2-sided [-0.025 to 0.082], Standard Error of Mean 0.027 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

11. Secondary Outcome: FVC AUC (0-6h) Response
Description: FVC AUC (0-6h) response [L] on day 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h, 4h, 5h, 6h after drug administration on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres | 0.283 (0.023) | 0.318 (0.024)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.2485, ANCOVA; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [-0.024 to 0.094], Standard Error of Mean 0.030 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

12. Secondary Outcome: FVC Peak 0-3h Response
Description: FVC peak 0-3h response [L] on day 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h after drug administration on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Number analyzed (Participants) | 136 | 136
Litres | 0.444 (0.033) | 0.490 (0.034)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio5 µg; Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.2875, ANCOVA; Mean Difference (Final Values) = 0.046, 95% CI 2-sided [-0.039 to 0.130], Standard Error of Mean 0.043 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

13. Secondary Outcome: PEFR AUC (0-3h) Response
Description: Peak Expiratory Flow Rate (PEFR) AUC (0-3h) response [L/min] on days 1, 15 and 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h after drug administration on days 1, 15 and 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres / minute
Groups:
- Olo 5 µg + Tio 5 µg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 136 | 136
Litres / minute
  Day 1 | 27.159 (1.604) | 28.143 (1.619)
  Day 15 | 27.817 (2.483) | 34.128 (2.507)
  Day 29 | 32.395 (2.101) | 33.947 (2.121)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.6299, ANCOVA; Mean Difference (Final Values) = 0.984, 95% CI 2-sided [-3.046 to 5.015], Standard Error of Mean 2.038 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.0475, ANCOVA; Mean Difference (Final Values) = 6.311, 95% CI 2-sided [0.070 to 12.553], Standard Error of Mean 3.156 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 3: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.5620, ANCOVA; Mean Difference (Final Values) = 1.552, 95% CI 2-sided [-3.729 to 6.833], Standard Error of Mean 2.670 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

14. Secondary Outcome: PEFR Peak 0-3h Response
Description: PEFR peak 0-3h response [L/min] on days 1, 15 and 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1h, 10min before drug administration and 5min, 30min, 1h, 2h, 3h after drug administration on days 1, 15 and 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres / minute
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 136 | 136
Litres / minute
  Day 1 | 49.125 (1.843) | 48.946 (1.861)
  Day 15 | 46.355 (2.801) | 52.835 (2.827)
  Day 29 | 52.497 (2.466) | 55.596 (2.490)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9391, ANCOVA; Mean Difference (Final Values) = -0.179, 95% CI 2-sided [-4.812 to 4.454], Standard Error of Mean 2.342 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.0709, ANCOVA; Mean Difference (Final Values) = 6.480, 95% CI 2-sided [-0.560 to 13.520], Standard Error of Mean 3.559 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 3: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.3245, ANCOVA; Mean Difference (Final Values) = 3.099, 95% CI 2-sided [-3.100 to 9.298], Standard Error of Mean 3.134 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

15. Secondary Outcome: PEFR AUC (6-12h) Response
Description: PEFR AUC (6-12h) response [L] on day 29.
  Response is defined as the change from baseline, baseline is defined as the mean of the 2 pre-treatment timepoints (-1 hour and -10 minutes) before first drug administration in each treatment period.
  The presented means are adjusted based on an ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed).
Time Frame: 1 hour (h) and 10 minutes before drug administration on day 1 and 6h, 9h and 12h after drug administration on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres / minute
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 130 | 132
Litres / minute | 24.830 (3.634) | 24.130 (3.599)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.8808, ANCOVA; Mean Difference (Final Values) = -0.700, 95% CI 2-sided [-9.914 to 8.514], Standard Error of Mean 4.655 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

16. Secondary Outcome: Weekly Mean Morning PEFR
Description: Weekly mean morning PEFR [L/min] on weeks 1,2,3 and 4.
  The presented means are adjusted.
Time Frame: Weeks 1,2,3 and 4
Population: FAS
Measure: Mean (Standard Error); unit: Litres / minute
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 131 | 132
Litres / minute
  Week 1 | 244.16 (1.713) | 245.28 (1.693)
  Week 2 | 242.38 (1.842) | 243.72 (1.821)
  Week 3 | 242.31 (1.805) | 242.97 (1.784)
  Week 4 | 242.90 (2.000) | 244.56 (1.977)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; Test week 1. Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.6081, ANCOVA; Mean Difference (Final Values) = 1.119, 95% CI 2-sided [-3.190 to 5.429], Standard Error of Mean 2.177 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; Test Week 2. Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.5686, ANCOVA; Mean Difference (Final Values) = 1.339, 95% CI 2-sided [-3.296 to 5.973], Standard Error of Mean 2.342 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 3: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; Test Week 3. Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.7765, ANCOVA; Mean Difference (Final Values) = 0.653, 95% CI 2-sided [-3.888 to 5.194], Standard Error of Mean 2.294 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 4: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; Test Week 4. Based on a ANCOVA with terms for baseline, treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.5166, ANCOVA; Mean Difference (Final Values) = 1.654, 95% CI 2-sided [-3.379 to 6.686], Standard Error of Mean 2.543 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

17. Secondary Outcome: Weekly Mean Evening PEFR
Description: Weekly mean evening PEFR [L/min] on weeks 1,2,3 and 4.
  The presented means are adjusted.
Time Frame: Weeks 1,2,3 and 4
Population: FAS
Measure: Mean (Standard Error); unit: Litres / minute
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 131 | 130
Litres / minute
  Week 1 | 262.21 (2.026) | 265.51 (2.024)
  Week 2 | 261.08 (2.146) | 262.47 (2.144)
  Week 3 | 258.62 (1.959) | 260.32 (1.956)
  Week 4 | 261.38 (1.942) | 260.34 (1.940)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.2037, ANCOVA; Mean Difference (Final Values) = 3.303, 95% CI 2-sided [-1.813 to 8.418], Standard Error of Mean 2.585 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 16, analysis 2]; Test type: Superiority or Other; p = 0.6118, ANCOVA; Mean Difference (Final Values) = 1.393, 95% CI 2-sided [-4.027 to 6.813], Standard Error of Mean 2.738 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 3: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 16, analysis 3]; Test type: Superiority or Other; p = 0.4988, ANCOVA; Mean Difference (Final Values) = 1.695, 95% CI 2-sided [-3.251 to 6.640], Standard Error of Mean 2.498 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 4: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 16, analysis 4]; Test type: Superiority or Other; p = 0.6757, ANCOVA; Mean Difference (Final Values) = -1.039, 95% CI 2-sided [-5.944 to 3.865], Standard Error of Mean 2.478 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

18. Secondary Outcome: Weekly Mean Number of Occasions of Rescue Therapy Used Per Day (PRN Salbutamol [Albuterol])
Description: Weekly mean number of occasions of rescue therapy used per day (as occasion require (PRN) salbutamol [albuterol]) on weeks 1,2,3 and 4.
  The means presented are the adjusted mean of weekly mean.
Time Frame: Weeks 1,2,3 and 4
Population: FAS
Measure: Mean (Standard Error); unit: number of occasions / day
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 131 | 132
number of occasions / day
  Week 1 | 1.294 (0.063) | 1.305 (0.062)
  Week 2 | 1.472 (0.068) | 1.352 (0.067)
  Week 3 | 1.369 (0.071) | 1.367 (0.070)
  Week 4 | 1.403 (0.071) | 1.363 (0.069)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.8901, ANCOVA; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.147 to 0.169], Standard Error of Mean 0.080 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 16, analysis 2]; Test type: Superiority or Other; p = 0.1647, ANCOVA; Mean Difference (Final Values) = -0.120, 95% CI 2-sided [-0.290 to 0.050], Standard Error of Mean 0.086 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 3: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 16, analysis 3]; Test type: Superiority or Other; p = 0.9822, ANCOVA; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.180 to 0.176], Standard Error of Mean 0.090 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 4: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 16, analysis 4]; Test type: Superiority or Other; p = 0.6542, ANCOVA; Mean Difference (Final Values) = -0.040, 95% CI 2-sided [-0.218 to 0.137], Standard Error of Mean 0.090 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

19. Secondary Outcome: Patient Global Rating
Description: Patient global rating scores treatment comparison after 4 weeks
  The score was evaluated on a 7-point scale :
  * 1 : very much better
  * 2 : much better
  * 3 : a little better
  * 4 : no change
  * 5 : a little worse
  * 6 : much worse
  * 7 : very much worse
  The presented means are adjusted.
Time Frame: 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 133 | 135
units on a scale | 3.207 (0.091) | 3.093 (0.090)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; Based on a ANCOVA with terms for treatment, centre, patient within centre and period (all effects fixed); Test type: Superiority or Other; p = 0.3269, ANCOVA; Mean Difference (Final Values) = -0.114, 95% CI 2-sided [-0.342 to 0.115], Standard Error of Mean 0.116 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

20. Secondary Outcome: Physician's Global Evaluation
Description: Physician's global evaluation score on days 15 and 29
  The score was evaluated on a 8-points scale :
  * Poor : 1,2
  * Fair : 3,4
  * Good : 5,6
  * Excellent : 7,8
  The presented means are adjusted
Time Frame: Days 15 and 29
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 135 | 136
units on a scale
  Day 15 | 5.084 (0.070) | 5.079 (0.070)
  Day 29 | 5.085 (0.063) | 5.065 (0.063)
Statistical Analysis 1: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.9557, ANCOVA; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.181 to 0.171], Standard Error of Mean 0.089 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg
Statistical Analysis 2: Comparison: Olo 2 µg + Tio 5 µg vs Olo 5 µg + Tio 5 µg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.8096, ANCOVA; Mean Difference (Final Values) = -0.019, 95% CI 2-sided [-0.178 to 0.140], Standard Error of Mean 0.080 — Difference calculated as Olo 5 µg + Tio 5 µg minus Olo 2 µg + Tio 5 µg

21. Secondary Outcome: Clinically Significant Abnormalities for Blood Chemistry, Haematology, Urinalysis and Physical Examination
Description: Clinically significant abnormalities for blood chemistry, haematology, urinalysis and physical examination
Time Frame: 14 weeks
Population: Treated Set (TS) including all randomized patients who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 138 | 138
participants
  Creatinine phosphokinase increased | 8 | 7
  Eosinophils increased | 3 | 3
  Urinalysis | 0 | 0

22. Secondary Outcome: Overall Marked Changes From Baseline in Vital Signs
Description: Overall marked changes from baseline in systolic blood pressure, diastolic blood pressure and pulse rate.
Time Frame: Baseline to week 14
Population: TS
Measure: Number; unit: participants
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 139 | 138
participants
  Systolic blood pressure increased | 16 | 23
  Systolic blood pressure decreased | 10 | 11
  Diastolic blood pressure increased | 19 | 15
  Diastolic blood pressure decreased | 13 | 17
  Pulse rate increased | 10 | 13
  Pulse rate decreased | 19 | 10

23. Secondary Outcome: 12-lead ECG Heart Rate
Description: 12-lead Electrocardiogram (ECG) Heart rate baseline and change from baseline values at other time points in Beats Per Minute (BPM)
  Statistics for each planned time from baseline to day 29.
Time Frame: Baseline, then 10min, 1h after drug administration on day 1, 30min before and 10min after drug administration on day 15, in addition 1h after drug administration on day 29
Population: TS
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 139 | 138
BPM
  Baseline | 72.96 (12.86) | 72.38 (11.96)
  Day1 0:10 | -1.44 (6.04) | -1.01 (5.63)
  Day1 1:00 | -2.09 (7.6) | -1.6 (7.45)
  Day15 -0:30 (N=137, 137) | 0.42 (11.09) | 1.1 (8.88)
  Day15 0:10 (N=135, 136) | -1.61 (8.77) | -0.79 (8.97)
  Day29 -0:30 (N=134, 136) | -0.69 (8.71) | 1.68 (9.43)
  Day29 0:10 (N=132, 135) | -2.14 (9.25) | -0.24 (9.5)
  Day29 1:00 (N=132, 135) | -2.34 (9.75) | -0.73 (8.98)

24. Secondary Outcome: 12-lead ECG PR Intervals
Description: 12-lead ECG PR intervals baseline and change from baseline at other timepoints in milliseconds.
  Statistics for each planned time from baseline to day 29.
Time Frame: as for outcome 23
Population: TS
Measure: Mean (Standard Deviation); unit: mS
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 139 | 138
mS
  Baseline | 160.03 (24.94) | 160.69 (29.28)
  Day1 0:10 | -1.02 (12.05) | -1.86 (17.53)
  Day1 1:00 (N=139, 137) | 2.12 (13.94) | 0.09 (11.07)
  Day15 -0:30 (N=136, 137) | 0.55 (12.56) | -0.95 (20.17)
  Day15 0:10 (N=135, 136) | 0.28 (12.17) | -1.24 (15.08)
  Day29 -0:30 (N=134, 135) | -1.29 (13.45) | -0.19 (15.35)
  Day29 0:10 (N=132, 135) | -0.29 (13.9) | -2.05 (16.39)
  Day29 1:00 (N=132, 135) | 1.98 (17.91) | 0.22 (13.05)

25. Secondary Outcome: 12-lead ECG QRS Intervals
Description: 12-lead ECG QRS intervals baseline and change from baseline at other time points in milliseconds
  Statistics for each planned time from baseline to day 29.
Time Frame: as for outcome 23
Population: TS
Measure: Mean (Standard Deviation); unit: mS
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 139 | 138
mS
  Baseline | 92.71 (11.92) | 92.41 (12.14)
  Day1 0:10 | -0.28 (6.29) | -0.65 (6.63)
  Day1 1:00 | -0.47 (6.39) | 0.31 (6.34)
  Day15 -0:30 (N=137, 137) | -0.55 (7.48) | -0.44 (7.73)
  Day15 0:10 (N=135, 136) | -0.67 (6.73) | -0.32 (7.9)
  Day29 -0:30 (N=134, 136) | -0.44 (7.55) | -0.75 (7.4)
  Day29 0:10 (N=132, 135) | -1.27 (6.63) | -0.82 (7.16)
  Day29 1:00 (N=132, 135) | -0.33 (7.5) | -0.39 (7.9)

26. Secondary Outcome: 12-lead ECG QTcF Intervals
Description: 12-lead ECG corrected heart rate (QT) interval, using Fridericia method (QTcF), baseline and change from baseline at other time points in milliseconds.
  Statistics for each planned time from baseline to day 29.
Time Frame: as for outcome 23
Population: TS
Measure: Mean (Standard Deviation); unit: mS
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 139 | 138
mS
  Baseline | 405.63 (21.42) | 403.53 (20.49)
  Day1 0:10 | -0.89 (12.85) | 0.97 (13.49)
  Day1 1:00 (N=138, 138) | -0.69 (12.79) | -0.61 (15.19)
  Day15 -0:30 (N=137, 137) | 0.55 (14.28) | -0.03 (16.5)
  Day15 0:10 (N=135, 136) | -1.16 (16.67) | -1.02 (17.37)
  Day29 -0:30 (N=134, 136) | -1.35 (17.18) | -0.24 (17.39)
  Day29 0:10 (N=132, 135) | -1.22 (15.05) | -2.08 (16.56)
  Day29 1:00 (N=132, 135) | -0.56 (18.24) | -1.05 (16.49)

27. Secondary Outcome: 12-lead ECG QTcB Intervals
Description: 12-lead ECG heart rate corrected QT interval, using Bazett method (QTcB), baseline and change from baseline at other time points in milliseconds.
  Statistics for each planned time from baseline to day 29.
Time Frame: as for outcome 23
Population: TS
Measure: Mean (Standard Deviation); unit: mS
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 139 | 138
mS
  Baseline | 418.12 (24.67) | 415.56 (23.35)
  Day1 0:10 | -2.18 (16.32) | 0.05 (16.14)
  Day1 1:00 (N=138, 138) | -2.57 (15.95) | -2.2 (18.05)
  Day15 -0:30 (N=137, 137) | 0.93 (18.23) | 0.91 (19.72)
  Day15 0:10 (N=135, 136) | -2.51 (20.37) | -1.76 (20.51)
  Day29 -0:30 (N=134, 136) | -1.87 (20.43) | 1.43 (21.52)
  Day29 0:10 (N=132, 135) | -3.13 (19.45) | -2.33 (20.35)
  Day29 1:00 (N=132, 135) | -2.55 (23.88) | -1.69 (19.75)

28. Secondary Outcome: 12-lead ECG QT Intervals
Description: 12-lead ECG QT intervals baseline and change from baseline at other time points in milliseconds.
  Statistics for each planned time from baseline to day 29.
Time Frame: as for outcome 23
Population: TS
Measure: Mean (Standard Deviation); unit: mS
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 139 | 138
mS
  Baseline | 382.73 (31.87) | 381.33 (29.42)
  Day1 0:10 | 1.59 (13.09) | 2.69 (13.82)
  Day1 1:00 (N=138, 138) | 2.97 (15.89) | 2.33 (18.02)
  Day15 -0:30 (N=137, 137) | -0.09 (19.95) | -1.76 (20.16)
  Day15 0:10 (N=135, 136) | 1.44 (20.59) | 0.53 (21.28)
  Day29 -0:30 (N=134, 136) | -0.59 (20.91) | -3.14 (20.13)
  Day29 0:10 (N=132, 135) | 2.27 (19.24) | -1.73 (20.83)
  Day29 1:00 (N=132, 135) | 3.14 (19.28) | 0.2 (20.51)

29. Secondary Outcome: AUC (0-6H) FEV1 (Unsupervised), AUC (0-6H) PEFR (Unsupervised), FVC Peak (0-3h), AUC (6-12h) FEV1 (Unsupervised), AUC (6-12h) PEFR (Unsupervised), Individual PEFR Measurements (Supervised and Unsupervised), Individual PEFR Measurements (Unsupervised)
Description: * AUC (0-6h) for FEV1, and PEFR (unsupervised) after first dose and after 2 and 4 weeks of treatment were not analysed in the study report because the pertinent information from the unsupervised Pulmonary Function Tests (PFTs) was for the time interval from 6 to 12 hours post-dosing.
  * FVC peak 0-3h response after the first dose and at Week 2 (supervised) and AUC (6-12h) for FEV1 and PEFR after the first dose and at Week 2 (unsupervised) were not analysed in the study report.
  * Individual PEFR (supervised) measurements and individual FEV1 and PEFR (unsupervised) measurements at each time point were not analysed in the study report.
Time Frame: 4 weeks
Population: No patients analyzed in the study report.
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio 5 µg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From drug administration until 14 days after the last administration, up to 12 weeks.
Arm/Group | Olo 2 µg + Tio 5 µg | Olo 5 µg + Tio5 µg
Serious Adverse Events (participants affected / at risk) | 3/139 | 5/138
Other Adverse Events (participants affected / at risk) | 23/139 | 16/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olo 2 µg + Tio 5 µg (N=139) | Olo 5 µg + Tio5 µg (N=138)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olo 2 µg + Tio 5 µg (N=139) | Olo 5 µg + Tio5 µg (N=138)
Nasopharyngitis (Infections and infestations) | 15 | 10
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.